CLINICAL TRIAL: NCT02946814
Title: Immediate Effect and Substantivity of the Essential Oils Without Alcohol on the Oral Biofilm in Situ. A Randomized Clinical Trial
Brief Title: Immediate Effect and Substantivity of the Essential Oils Without Alcohol on the Oral Biofilm in Situ
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Inmaculada Tomas, Senior Lecturer, University of Santiago de Compostela
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: substantivity 2016
Record Dates: First submitted 2016-10-21; First posted 2016-10-27 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Biofilms; Substantivity; Oils, Essential
Keywords: essential oils; microscope, colfocal; dental plaque
MeSH Terms: conditions — Dental Plaque | interventions — Oils, Volatile; Mouthwashes

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- essential oils (Active Comparator): a single mouthwash with 20 ml of essential oils for 30 seconds.
  Interventions: Drug: essential oils
- essential oils without mouthwash (Experimental): a single mouthwash with 20 ml of essential oils without alcohol for 30 seconds.
  Interventions: Drug: essential oils without mouthwash
- sterile water (Sham Comparator): a single mouthwash with 20 ml of sterile water for 30 seconds.
  Interventions: Drug: sterile water

INTERVENTIONS:
Drug: essential oils
  Other Names: Listerine Mentol
  Arms: essential oils
Drug: essential oils without mouthwash
  Other Names: Listerine Zero
  Arms: essential oils without mouthwash
Drug: sterile water
  Arms: sterile water

SUMMARY:
This study aims to evaluate the in situ antibacterial activity of a mouthwash containing essential oils with and without alcohol on undisturbed de novo plaque-like biofilm (PL-biofilm) up to 7 h after its application.

An appliance was designed to hold six glass disks on the buccal sides of the lower teeth, allowing PL-biofilm growth. Twenty healthy volunteers will the appliance for 48 h and then performed a mouthwash with essential oils. Disks will be removed after 30 s and at 1, 3, 5, and 7 h later. After a washout period, the same procedure will be repeated with a sterile water mouthwash and a mouthwash with essential oils without alcohol. After PL-biofilm vital staining, samples will be analyzed using a confocal laser scanning microscope analysing their bacterial viability and thickness.

ELIGIBILITY:
Inclusion Criteria:

Systemically healthy adults.

* Minimum of 24 permanent teeth.
* No gingivitis (Community Periodontal Index score = 0).
* No periodontitis (Community Periodontal Index score = 0).
* Absence of untreated caries.

Exclusion Criteria:

* Smoker or former smoker.
* Presence of dental prostheses.
* Presence of orthodontic devices.
* Antibiotic treatment or routine use of oral antiseptics in the previous 3 months.
* Presence of any systemic disease that could alter the production or composition of saliva.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-10; Primary Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of bacterial viability | 48 hours after the volunteer has started to wear the splints

SECONDARY OUTCOMES:
thickness in microns | 48 hours after the volunteer has started to wear the splints

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quintas V, Prada-Lopez I, Prados-Frutos JC, Tomas I. In situ antimicrobial activity on oral biofilm: essential oils vs. 0.2 % chlorhexidine. Clin Oral Investig. 2015 Jan;19(1):97-107. doi: 10.1007/s00784-014-1224-3. Epub 2014 Apr 1. PMID 24687247